CLINICAL TRIAL: NCT05738876
Title: Non Obstructive Versus Obstructive Coronary Artery Disease Documented by Coronary Angiography; Prevalence & Diagnostic Features in a Single Center Experience : A Prospective Cross Sectional Study
Brief Title: Non Obstructive Versus Obstructive Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Arab Board of Health Specializations, Iraq (Other)
Responsible Party: Principal Investigator, Hasanain Ali Al ftailah, Non obstructive versus obstructive coronary artery disease documented by coronary angiography; prevalence & diagnostic features in a single center experience : A prospective cross sectional study, Arab Board of Health Specializations, Iraq
Other Study IDs: NOCAD diagnostic features
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Non-Obstructive Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CORONARY ANGIOGRAPHY — coronary angiography by femoral or radial artery access

SUMMARY:
The goal of this observational study is to study the non obstructive type of ischemic heart disease by identifying unique clinical features , frequency and age group .in patient admitted in coronary care unit , suffered from angina or heart attack. . The main question[s] it aims to answer are:

* how it different from classical type of ischemic heart disease ( obstructive coronary artery disease)
* what is frequency and age prevalence of these patient Participants evaluated by history , clinical examination, serum troponin and coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IHD ( MI, unstable angina ,chronic stable angina)
* >18 years of age
* patients undergoing CAG for emergency or elective situations.

Exclusion Criteria:

* Patients who were hemodynamically unstable.
* patients with incomplete data
* patients with clinical features of pericarditis or others of non cardiac origin chest pain .

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with clinical features of IHD underwent coronary angiography in CCU of imam hussain hospital from January to May of 2021
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Non obstructive versus obstructive coronary artery disease documented by coronary angiography; prevalence & diagnostic features in a single center experience : A prospective cross sectional study | BASELINE
  analysis of diagnostic features and frequency of non obstructive artery disease in comparison to obstructive artery disease

CONTACTS AND LOCATIONS:
Locations (1):
- Arab board of health specializations-Iraq, Karbala , Iraq, Karbala, Iraq